CLINICAL TRIAL: NCT02946450
Title: Multi-center, Prospective, Non-interventional, Observational Study to Assess the Safety of Omnipure® Inj.(Iohexol) Contrast Media in CT Scanning Patients
Brief Title: Observational Study to Assess the Safety of Omnipure® Inj.(Iohexol) Contrast Media in CT Scanning Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_IOH001
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: CT Scanning Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Not applicable-observational study: Not applicable-observational study
  Interventions: Drug: Other: Not applicable-observational study

INTERVENTIONS:
Drug: Other: Not applicable-observational study

SUMMARY:
The purpose of this study is to assess safety of Omnipure inj. (lohexol) contrast media in CT scanning patients

ELIGIBILITY:
Inclusion Criteria:

* subjects in need of CT scanning
* subjects who signed up informed consent

Exclusion Criteria:

* Known allergy or hypersensitivity to the study medication, ingredient of the medication, and Iodine type medication
* severe renal insufficiency patients
* severe hypothyroidism
* severe local infection or bacteremia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CT scanning patients
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
adverse events, adverse drug reaction, serious adverse events, serious drug reaction, laboratory data, vital signs | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No